CLINICAL TRIAL: NCT00675129
Title: A Randomized Controlled Trial for Repetitive Deliberate Self-harm and Suicidal Behaviours Among Norwegian Adolescents: a Comparison Between Dialectical Behaviour Therapy Adapted for Adolescents (DBT-A) and Enhanced Usual Care (EUC)
Brief Title: Treatment for Adolescents With Deliberate Self Harm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Mehlum, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHDIR-04-627
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Intentional Self Harm
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Therapeutics; Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dialectical behavioral therapy
  Interventions: Behavioral: Dialectical behavioral therapy for adolescents (DBT-A)
- 2 (Active Comparator): Enhanced Usual Care (standard care plus monitoring and patient safety protocol implemented)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy for adolescents (DBT-A) — Patients randomised to DBT-A will receive 16 weeks treatment, with one weekly session (60 minutes)of individual therapy, one weekly session of multifamily skills training (120 minutes), and telephone coaching outside therapy sessions.
  The treatment has been developed by Marsha Linehan (Linehan, 1993a; 1993b)and adapted for adolescents by Alec Miller (Miller, Rathus & Linehan, 2007). Individual DBT therapists have been trained by drs Alec L Miller and Sarah K Reynolds and have a minimum of one year clinical practise as DBT therapists. The therapists are organised in two consultation teams supervised on a bimonthly basis throughout the entire study by drs Miller and Reynolds respectively.
  Arms: 1
Behavioral: Treatment as usual — Patients randomised to EUC will received standard care (16 weeks) at five participating child and adolescent outpatient clinics from therapists not trained in or practising DBT. According to pilot study data EUC will most likely consist of psychodynamic therapy, various forms of family therapy and supportive therapy.
  Other Names: Psychosocial intervention
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the efficiency of dialectical behavior therapy (DBT) in treatment of adolescents with deliberate self harm compared to Enhanced Usual Care (EUC). Eighty patients in the age of 12-18 yrs old will be included in the study. The main inclusion criterion is repetitive deliberate self-harm. The patients will receive 16 weeks treatment in outpatient clinics in Oslo, after having been randomized to DBT or EUC. They will be assessed on five different time-points: baseline (before starting treatment), 6 weeks (after start of treatment), 12 weeks, 16 weeks and 68 weeks.

The main study hypothesis is:

* DBT will be significantly more effective in treatment of self-harm behavior, as measured/indicated by reduction in number of self-harm episodes with or without intent to die, as well as reduction of number of emergency room visits.
* It is also hypothesized that DBT will significantly reduce the level of suicidal ideation and depressive symptoms compared to EUC.

DETAILED DESCRIPTION:
Power analysis:

Exact data on the repetition of self-harm over 16-20 week and 12 months observation periods for adolescents in outpatient psychiatric treatment are not available. Building on previous clinical studies and RCT studies in adults receiving DBT, we anticipate that the 16 week repetition rate will be 50% for adolescents who receive EUC and 25% for adolescents who receive DBT. With an alpha error level of 5% 60 patients in each group is needed to provide 80% power with a two tailed test. We anticipate a drop out rate from research assessments of no more than 25%. To compensate for this attrition, it is calculated that 15 patients in each treatment group should be added, leading to a total number of 150 patients to be included in the trial. A more precise power analysis and determination of how many patients to include in the study will be based on data from the first 40 patients who have been included.

A power analysis conducted on the basis of the first 40 patients showed that:

1. There had been no attrition from research assessments
2. With an alpha error level of 5% 40 patients in each group is needed to provide 80% power with a two tailed test

A final number of patients to include was therefore fixed at 80.

ELIGIBILITY:
Inclusion Criteria:

* History of repeated deliberate self harm (last episode within last months)
* Satisfies at least 2 criteria of DSM-IV Borderline Personality Disorder (as measured by SCID-II) in addition to the self-destructive criterion.

Or: Satisfies at least 1 criterion + 2 criteria scored below threshold (score 2) of DSM-IV Borderline Personality Disorder (as measured by SCID-II) in addition to the self-destructive criterion.

Exclusion Criteria:

* Psychotic disorders
* Anorexia Nervosa
* Substance dependence disorder
* Mental retardation (IQ less than 70)
* Asperger syndrome/autism

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2008-05; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Frequency of subsequent episodes of deliberate self harm and time elapsed to future episodes of deliberate self harm | 16 weeks and 68 weeks
Severity of suicidal ideation, level of depressive symptoms | 16 weeks and 68 weeks

SECONDARY OUTCOMES:
Frequency of subsequent emergency room visits, hospitalizations and use of additional treatments due to risk of deliberate self-harm behavior | 16 weeks and 68 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Mehlum, Professor, Principal Investigator — Suicide Research and Prevention Unit/University of Oslo
Locations (1):
- Suicide Research and Prevention Unit/University of Oslo, Oslo, Norway

REFERENCES:
- [Background] Linehan, M.M. (1993a). Cognitive-behavioral treatment of borderline personality disorder. New York: Guilford Press
- [Background] Linehan, M.M. (1993b). Skills training manual for treating borderline personality disorder. New York: Guilford Press
- [Background] Miller, A.L., Rathus J.H., Linehan, M.M. (2007). Dialectical behavioral therapy with suicidal adolescents. New York: Guilford Press
- [Derived] Dibaj IS, Tormoen AJ, Klungsoyr O, Morken KTE, Haga E, Dymbe KJ, Mehlum L. Early remission of deliberate self-harm predicts emotion regulation capacity in adulthood: 12.4 years follow-up of a randomized controlled trial of adolescents with repeated self-harm and borderline features. Eur Child Adolesc Psychiatry. 2025 Jun;34(6):1837-1848. doi: 10.1007/s00787-024-02602-8. Epub 2024 Oct 29. PMID 39470788
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Ramleth RK, Groholt B, Diep LM, Walby FA, Mehlum L. The impact of borderline personality disorder and sub-threshold borderline personality disorder on the course of self-reported and clinician-rated depression in self-harming adolescents. Borderline Personal Disord Emot Dysregul. 2017 Oct 31;4:22. doi: 10.1186/s40479-017-0073-5. eCollection 2017. PMID 29093819
- [Derived] Mehlum L, Ramberg M, Tormoen AJ, Haga E, Diep LM, Stanley BH, Miller AL, Sund AM, Groholt B. Dialectical Behavior Therapy Compared With Enhanced Usual Care for Adolescents With Repeated Suicidal and Self-Harming Behavior: Outcomes Over a One-Year Follow-Up. J Am Acad Child Adolesc Psychiatry. 2016 Apr;55(4):295-300. doi: 10.1016/j.jaac.2016.01.005. Epub 2016 Jan 27. PMID 27015720
- [Derived] Mehlum L, Tormoen AJ, Ramberg M, Haga E, Diep LM, Laberg S, Larsson BS, Stanley BH, Miller AL, Sund AM, Groholt B. Dialectical behavior therapy for adolescents with repeated suicidal and self-harming behavior: a randomized trial. J Am Acad Child Adolesc Psychiatry. 2014 Oct;53(10):1082-91. doi: 10.1016/j.jaac.2014.07.003. Epub 2014 Jul 22. PMID 25245352
- See also: Information about the research project in Norwegian — http://www.med.uio.no/ipsy/ssff/forskning/dbt/forskningsprosjekt_dbt.html
- See also: The Suicide Research and Prevention Unit/University of Oslo - information in English — http://www.med.uio.no/ipsy/ssff/english/index_english.html